CLINICAL TRIAL: NCT06481059
Title: Soluble Urokinase Plasminogen Activator Receptor (suPAR) is a Potential Biomarker of Stage III-IV, Grade C Periodontitis Through the Impact of Post-radiotherapy on Head and Neck Cancer Patients
Brief Title: suPAR is a Potential Biomarker of in Chronic Periodontitis Through the Impact of Post-radiotherapy on HNCs Patients
Acronym: HNCs
Status: Completed | Type: Observational
Sponsor: Al-Maarif University College (Other)
Responsible Party: Sponsor
Other Study IDs: suPAR as a biomarker
Record Dates: First submitted 2024-06-22; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Head and Neck Cancer; Chronic Periodontitis; Radiotherapy; Complications
MeSH Terms: conditions — Head and Neck Neoplasms; Chronic Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head and neck cancer post-radiotherapy: Head and neck cancer patients who received radiotherapy after six months. fractions no. [(32-35 fractions) 5700-7000 Gy] addition chemotherapy [(cisplatin or cetuximab) (2-3 doses)].
  Interventions: Radiation: Head and Neck cancer post-radiotherapy

INTERVENTIONS:
Radiation: Head and Neck cancer post-radiotherapy — Head and Neck Cancer patients who received radiotherapy after 6 months
  Other Names: Head and neck cancer patients after 6 irradiation

SUMMARY:
This study aims to improve a soluble urokinase plasminogen activator receptor suPAR is a reliable biomarker of chronic periodontitis and may be replaced in patients with head and neck cancer post-radiotherapy (HNC post-RT).

DETAILED DESCRIPTION:
The urokinase-type plasminogen activator receptor (uPAR) plays an essential function in leukocytes and endothelial homeostasis and, therefore, in the development of chronic periodontitis. The study enrolled 150 participants, 50 chronic periodontitis with head and neck cancer post radiotherapy (CP+HNC post-RT) patients, 50 chronic periodontitis (CP) without HNC patients, and 50 healthy controls. Clinical Attachment Loss (CAL), Probing Pocket Depth (PPD), Plaque Index (PI), and Gingival Bleeding Index (GBI) were recorded. An enzyme-linked immunosorbent assay (ELISA) was constructed to quantify serum (suPAR) levels. Stage and grade of periodontitis were stage III-IV, grade C in patients (CP+HNC post-RT), stage I-III, grade A/B in patients (CP without HNC), and absent in (healthy). Chronic periodontitis with HNC post-RT patients presented a significantly higher proportion of suPAR levels (506.7 pg/ml) compared to chronic periodontitis without HNC and healthy controls (423.08 pg/ml and 255.9 pg/ml), respectively. A significant positive correlation was found between serum suPAR levels and CAL, PPD, PI, and GBI in the periodontal disease groups. ROC results of suPAR (AUC=0.976 for CP+HNC post-RT, AUC=0.872 for CP without HNC). Hyposalivation appeared in patients (CP+HNC post-RT; 0.15 [0.11-0.23] ml/min, P=0.001) and (CP without HNC; 0.30 [0.25-0.41] ml/min, P=0.001), compared to healthy controls; 0.35 [0.28- 0.54] ml/min, P=0.001). The study showed a significant elevation in serum suPAR levels in CP+HNC post-RT patients compared to the CP without HNC and control groups.

ELIGIBILITY:
Inclusion Criteria:

* A pathologically confirmed malignant neoplasm of HNC (derived from epithelial cells).
* Not having received radiation therapy previously.
* No distant metastasis.
* No history of salivary gland surgery (parotid, submandibular, or sublingual).
* A generally satisfactory physical condition with a performance score of 0 to 1 point and a planned survival period of more than a year and scores of 2 higher indicating increasing disability.

Exclusion Criteria:

* Previous oral disease or salivary gland disease history.
* Definitive diagnosis of multiple sclerosis, xerostomia, or systemic disease.
* Refusal to participate in the study.

Ages: 28 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was n=26 nasopharyngeal tumors (n=20 nonkeratinizing and n=6 keratinizing carcinomas), (n=6 oropharyngeal squamous cell carcinoma, SCC), (n=8 Laryngeal cancer), (n=6 tongue cancer), and (n=4 primary malignancies of unclear origin). Many patients had a history of smoking, and the mean patient age was 45.8 years (min-max: 28-72 years); 40 (80%) were men. Twenty-eight of the patients (or 56%) had a concomitant systemic therapy (2-3 doses) of cisplatin or cetuximab in addition to radiotherapy. Chronic periodontitis patients (n=50) without HNCs. More than half of them had a history of smoking, with 31 (62%) and 5 (10) of them having used alcohol. A control group (n=50) was used periodontally healthy.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Measure of serum suPAR level | at 6 months
  Measure of serum suPAR level in patients head and neck cancer who received radiotherapy

SECONDARY OUTCOMES:
Periodontal parameters measured | at 6 month
  All periodontal parameters (Clinical attachment level, Gingival bleeding Index, Plaque index, and Periodontal pocket depth measures were performed manually using a millimeter periodontal probe in patients who received radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A. Al-Kubaisi, PhD, Study Director — Al-Maarif University College; Maysam A. Ghazi, MSc, Study Chair — Al-Maarif University College; Nisreen S. Majeed, MSc, Study Chair — Al-Maarif University College; Ekram R. Aldelaimi, BDS, Study Chair — Department of Periodontology, Al-Anbar Health Directorate, Ministry of Health; Hamid H. Enezei, PhD, Study Director — Department of Oral and Maxillofacial Surgery, College of Dentistry, University of Anbar
Locations (1):
- Ahmed A. Al-Kubaisi, Ramadi, Al-Anbar Governorate, Iraq

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gasparoni LM, Alves FA, Holzhausen M, Pannuti CM, Serpa MS. Periodontitis as a risk factor for head and neck cancer. Med Oral Patol Oral Cir Bucal. 2021 Jul 1;26(4):e430-e436. doi: 10.4317/medoral.24270. PMID 33340075
- [Result] Lalla RV, Treister NS, Sollecito TP, Schmidt BL, Patton LL, Helgeson ES, Lin A, Rybczyk C, Dowsett R, Hegde U, Boyd TS, Duplinsky TG, Brennan MT. Radiation therapy for head and neck cancer leads to gingival recession associated with dental caries. Oral Surg Oral Med Oral Pathol Oral Radiol. 2022 May;133(5):539-546. doi: 10.1016/j.oooo.2022.01.016. Epub 2022 Jan 31. PMID 35304084